CLINICAL TRIAL: NCT00376467
Title: STI 571 (GLIVEC) in the Treatment of Philadelphia-chromosome Positive and/or BCR/ABL Rearranged Adult Acute Lymphoblastic Leukemia. GIMEMA LAL 0201.
Brief Title: STI 571 (GLIVEC) in the Treatment of Adult Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL0201
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Philadelphia positive; Adult; Elderly; Imatinib
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib

SUMMARY:
This proposal, developed in the framework of the GIMEMA, will permit:

* to evaluate the activity and toxicity of imatinib in the treatment of Ph+ acute lymphoblastic leukemia;
* to evaluate the molecular response to the treatment, and to monitor the molecular status of remission in all cases achieving or not a molecular response.

The GIMEMA has activated a network to centralize all biological samples (bone marrow and peripheral blood) at diagnosis from all new ALL patients. This will permit to identify, in particular, Ph + and/or BCR/ABL + cases within 5 days from diagnosis, thus permitting to treat these patients according to different programs on the basis of the presence of Ph chromosome.

DETAILED DESCRIPTION:
Imatinib shows a specific activity for the ABL protein- tyrosine kinase at the in vitro and in vivo level. The compound exerts a direct inhibition on the proliferation of BCR/ABL+ve cells, in cell lines derived from ALL and CML patients, inducing apoptosis. Induction of apoptosis by imatinib was observed also in primary samples of leukemic cells obtained from Ph+ve ALL patients. Since activated BCR/ABL tyrosine kinase is present in nearly all patients with CML and in 25-30% of those with ALL, these two diseases are the ideal targets to verify the potential therapeutic activity of this ABL specific tyrosine kinase inhibitor. So far only limited experiences on the therapeutic benefit of imatinib in ALL patients have been referred. In one of these studies, all 10 treated patients had received prior chemotherapeutic treatment for their leukemia. Imatinib was administered as daily oral therapy and all patients were treated on outpatient basis. Different dosages were tested: 300, 400, 500 mg/day for 28 days. Some responding patients showed prolonged myelosuppression, but only a minority of these required hospitalization, while other side effects appeared acceptable. Although these results demonstrated that Imatinib, as a single agent, is active in BCR/ABL +ve ALL, being able to induce a high response rate, however these responses appeared to be short. This occurred mainly in patients with advanced leukemia, thus it could be hypothesized that early relapse, in these patients, may due to a pre-existing resistance or developed resistance to Imatinib. In vitro studies as well as limited preclinical experiences are showing enhanced antileukemic effects of Imatinib in combination with cytotoxic drugs, thus further clinical trials should be aimed to ascertain, mainly in previously untreated patients, which are the optimal dosage and the best duration of treatment for maximal therapeutic benefit and to test if this agent, combined with conventional chemotherapy, could really enhance its antileukemic activity.

The Gimema Group will run two distinct studies among the same protocol to verify the antileukemic activity and safety of imatinib in Ph+ve and/or BCR/ABL +ve ALL:

Study A: Imatinib as post-consolidation therapy in adult (>=18 and <=60 yrs) ALL patients in 1st CHR; Study B: Imatinib without chemotherapy for remission induction in elderly (>60 years) ALL patients.

This proposal, developed in the framework of the GIMEMA, will include:

1. centralization of all biological samples (bone marrow and peripheral blood) at diagnosis from all new ALL patients, to identify, in particular, Ph + and/or BCR/ABL + cases;
2. evaluation of the molecular response to the treatment, and monitoring the molecular status during the hematological remission in all cases in CR;
3. treatment of all adult patients with the same induction and consolidation treatment already used in the past by GIMEMA for Ph+ ALL, to have also the possibility of an historical control versus patients treated before the "imatinib era".

Study A: Imatinib in Ph +ve and/or BCR/ABL +ve adult (age <60 years) ALL patients in first CHR after induction and consolidation treatment.

Aimed to verify the activity and safety of STI 571 administered after the induction and consolidation therapy in Ph+ve and/or Bcr/Abl+ve ALL patients in 1st CHR (+CMR). A cohort of 38 patients will be enrolled. All Gimema Centers can join this study. Quantitative Rt-PCR assay is mandatory before start of Imatinib treatment.

Patients will receive on an out-patients basis Imatinib p.o. at the dosage of 400 mg x 2/daily for 6 months. After completing the 6-months therapy, and in absence of safety concerns, patients may receive additional therapy with Imatinib, provided that, in the opinion of investigator, the patient has benefited from treatment.

Study B: Imatinib as induction treatment in newly diagnosed Ph+ and/or Bcr/Abl+ elderly (age >60 years) ALL patients.

Aimed to verify the activity and safety of Imatinib combined with steroids during the induction phase in elderly (>60 years) Ph+ve and/or Bcr/Abl+ve ALL patients. A cohort of 53 patients will be enrolled. All Gimema Centers can join this study. The cytogenetic and/or molecular diagnosis must be obtained within 5 days from diagnosis.

Patients will receive Imatinib p.o at the dosage of 400 mg x 2/daily for 30 days on an out-patients basis. After completing induction therapy patients may receive additional therapy with Imatinib, provided that, in the opinion of investigator, the patient benefited from treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ph +ve and/or BCR/ABL +ve ALL, either in 1st CHR (independently from the molecular status) for study A, or at diagnosis and untreated for study B;
* Age >18 years and <60 for study A, >60 for study B;
* Written voluntary informed consent.

Exclusion Criteria:

* Patients of childbearing potential without a negative pregnancy test prior to the initiation of study. Barrier contraceptive precautions are to be used throughout the trial in both sexes;
* Pretreatment with steroids for more than 10 days in study B;
* Serum bilirubin and creatinine values >3 the upper limit of normal range;
* SGOT and SGPT values >3 the upper limit of the normal range;
* Patients who had received any other investigational agent within 4 weeks before the enrollment;
* Patients with cardiovascular diseases grade >3 according to the New York Heart Association (see Appendix 1);
* Patients with a history of non compliance to medical regimen or who are considered potentially unreliable;
* Patients with moderate/severe mood or psychiatric disorders;
* Concomitant neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-12; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
for Study A, the primary endpoint for activity is overall CMR rate | after 6 months of imatinib treatment
for Study B, the primary endpoint for activity is overall CHR (+/- CMR) rate . | after induction treatment

SECONDARY OUTCOMES:
complete hematological or molecular remission duration | at study end
overall survival. | at study end

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, Principal Investigator — Università degli Studi di Udine
Locations (28):
- Italy (28):
  - Divisione di Ematologia, Azienda Policlinico "Umberto I", Università degli Studi "La Sapienza", Rome, Rome
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - Az.Ospedaliera S.G.Moscati, Avellino
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Ferrara
  - Ospedale Niguarda " Ca Granda", Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologi, Modena
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Servizio Sanitario Nazionale - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli" - Struttura Complessa di Ematologia - Div. TERE- 4° piano - Padiglione Palermo, Napoli
  - zienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - U.O. di Oncoematologia di Nocera Inferiore-plesso ospedaliero "A. Tortora" di Pagani del DEA Nocera-Pagani, Nocera Inferiore
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2, Orbassano
  - La Maddalena Casa di Cura di Alta Specialità Dipartimento Oncologico di III Livello, Palermo
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Ematologia - Ospedale San Carlo, Potenza
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Azienda Sanitaria Locale Viterbo - Polo Ospedaliero Centrale - Ospedale Di Ronciglione - U.O. di Ematologia, Ronciglione
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, S. G. Rotondo
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

REFERENCES:
- [Result] Vignetti M, Fazi P, Cimino G, Martinelli G, Di Raimondo F, Ferrara F, Meloni G, Ambrosetti A, Quarta G, Pagano L, Rege-Cambrin G, Elia L, Bertieri R, Annino L, Foa R, Baccarani M, Mandelli F. Imatinib plus steroids induces complete remissions and prolonged survival in elderly Philadelphia chromosome-positive patients with acute lymphoblastic leukemia without additional chemotherapy: results of the Gruppo Italiano Malattie Ematologiche dell'Adulto (GIMEMA) LAL0201-B protocol. Blood. 2007 May 1;109(9):3676-8. doi: 10.1182/blood-2006-10-052746. Epub 2007 Jan 9. PMID 17213285